CLINICAL TRIAL: NCT03819920
Title: Does Knowing One's Estimated Colorectal Cancer Risk Influence Screening Behavior?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Uri Ladabaum, Professor of Medicine, Director GI Cancer Prevention Program, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-32815
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: cancer screening beliefs; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Risk Assessment

STUDY DESIGN:
Intervention Model Description: Usual care of generalized colorectal cancer screening education over telephone versus personalized risk assessment over telephone using National Cancer Institute Colorectal Cancer Risk Assessment Tool (CCRAT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (Placebo Comparator): Patients receive standardized general information about colorectal cancer screening over the telephone.
  Interventions: Behavioral: Usual Care (UC)
- Risk Assessment (CCRAT) (Active Comparator): Patient receive personalized colorectal cancer risk assessment over the telephone by answering the questions as outlined in the National Cancer Institute Colorectal Cancer Risk Assessment Tool (https://ccrisktool.cancer.gov/calculator.html)
  Interventions: Behavioral: Risk Assessment (CCRAT); Behavioral: Usual Care (UC)

INTERVENTIONS:
Behavioral: Risk Assessment (CCRAT) — Patient receive personalized colorectal cancer risk assessment over the telephone by answering the questions as outlined in the National Cancer Institute Colorectal Cancer Risk Assessment Tool (https://ccrisktool.cancer.gov/calculator.html)
  Other Names: CCRAT
  Arms: Risk Assessment (CCRAT)
Behavioral: Usual Care (UC) — Patients receive standardized general information about colorectal cancer screening over the telephone.
  Other Names: UC

SUMMARY:
This study is designed to examine the impact of telephone-based colorectal cancer risk assessment on colorectal screening attitudes and behavior among previously unscreened adults ages 50 to 75.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) remains the 3rd most common cancer in the US. Most CRCs are preventable, but screening participation remains suboptimal. Several factors have been associated with screening compliance, such as perception of CRC risk. Here we study the impact of telephone-based administration of the National Cancer Institute Colorectal Cancer Risk Assessment Tool (CCRAT) compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any participating physician
* Not having had any colorectal cancer screening test prior
* Able to speak English

Exclusion Criteria:

* Personal history of inflammatory bowel disease
* Personal history of colorectal cancer
* Personal history of Lynch syndrome or Familial Adenomatous Polyposis
* Have already received colorectal cancer screening

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Screening Behavior: Differences in colorectal cancer screening completion rates between usual care (UC) and CCRAT | 12 months after intervention
  Any CRC screening test completed including stool tests (FOBT (fecal occult blood test), FIT (immunochemical test for fecal blood), stool DNA test), colonoscopy, flexible sigmoidoscopy, double contrast barium enema, CT colonography (virtual colonoscopy)

SECONDARY OUTCOMES:
Screening Behavior: Differences in colorectal cancer screening completion rates between usual care (UC) and CCRAT | 6 months after intervention
  Any CRC screening test completed including stool tests (FOBT (fecal occult blood test), FIT (immunochemical test for fecal blood), stool DNA test), colonoscopy, flexible sigmoidoscopy, double contrast barium enema, CT colonography (virtual colonoscopy)
Change in intention to screen at 6 months and 12 months | Immediate after intervention, 6 months and 1 year after intervention
  Differences in progressive behavioral stages of adoption from precontemplation to contemplation to preparation.
Colorectal cancer screening rates at 12 months as a function of CCRAT score | 12 months after intervention
  Screening completion at 12 months will be compared between the 3 tertiles of CCRAT score in the intervention group to determine whether there is any relationship between absolute CCRAT score and screening completion

OTHER OUTCOMES:
Risk perception: Health Belief Model Likert Scale | Immediate after intervention
  Differences in perception of one's own risk of colorectal cancer ranging from "very unlikely" (minimum) to "very likely" (maximum), with "very unlikely" representing the most favorable outcome of perceived risk and "very likely" representing the most unfavorable outcome of perceived risk.
Fear: Health Belief Model Likert Scale | Immediate after intervention
  Presence of fear of discovering colorectal cancer on performing screening test ranging from "strongly disagree" (minimum) to "strongly agree" (maximum), with "strongly disagree" representing the most favorable outcome of fear and "strongly agree" representing the most unfavorable outcome of fear.

CONTACTS AND LOCATIONS:
Overall Officials: Uri Ladabaum, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made available to other researchers through a HIPAA compliant data storage system (Stanford Medicine Box) that is password protected
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2/1/2019-2/1/2021
Access Criteria: Research staff solely associated with the study and/or Graduate or Post-Doc students-who are writing related manuscripts - who have been given permission by the Principal Investigator, Uri Ladabaum can submit a request.

REFERENCES:
- [Background] Volk RJ, Linder SK, Lopez-Olivo MA, Kamath GR, Reuland DS, Saraykar SS, Leal VB, Pignone MP. Patient Decision Aids for Colorectal Cancer Screening: A Systematic Review and Meta-analysis. Am J Prev Med. 2016 Nov;51(5):779-791. doi: 10.1016/j.amepre.2016.06.022. Epub 2016 Sep 2. PMID 27593418
- [Background] Champion VL, Christy SM, Rakowski W, Gathirua-Mwangi WG, Tarver WL, Carter-Harris L, Cohee AA, Marley AR, Jessup NM, Biederman E, Kettler CD, Stump TE, Monahan P, Lairson DR, Rawl SM. A Randomized Trial to Compare a Tailored Web-Based Intervention and Tailored Phone Counseling to Usual Care for Increasing Colorectal Cancer Screening. Cancer Epidemiol Biomarkers Prev. 2018 Dec;27(12):1433-1441. doi: 10.1158/1055-9965.EPI-18-0180. Epub 2018 Sep 4. PMID 30181203
- [Background] Miller DP Jr, Denizard-Thompson N, Weaver KE, Case LD, Troyer JL, Spangler JG, Lawler D, Pignone MP. Effect of a Digital Health Intervention on Receipt of Colorectal Cancer Screening in Vulnerable Patients: A Randomized Controlled Trial. Ann Intern Med. 2018 Apr 17;168(8):550-557. doi: 10.7326/M17-2315. Epub 2018 Mar 13. PMID 29532054
- [Background] Christy SM, Rawl SM. Shared decision-making about colorectal cancer screening: a conceptual framework to guide research. Patient Educ Couns. 2013 Jun;91(3):310-7. doi: 10.1016/j.pec.2013.01.015. Epub 2013 Feb 15. PMID 23419327
- [Background] Schroy PC 3rd, Duhovic E, Chen CA, Heeren TC, Lopez W, Apodaca DL, Wong JB. Risk Stratification and Shared Decision Making for Colorectal Cancer Screening: A Randomized Controlled Trial. Med Decis Making. 2016 May;36(4):526-35. doi: 10.1177/0272989X15625622. Epub 2016 Jan 19. PMID 26785715
- [Background] Han PK, Duarte CW, Daggett S, Siewers A, Killam B, Smith KA, Freedman AN. Effects of personalized colorectal cancer risk information on laypersons' interest in colorectal cancer screening: The importance of individual differences. Patient Educ Couns. 2015 Oct;98(10):1280-6. doi: 10.1016/j.pec.2015.07.010. Epub 2015 Jul 19. PMID 26227576
- [Background] Vernon SW, Bartholomew LK, McQueen A, Bettencourt JL, Greisinger A, Coan SP, Lairson D, Chan W, Hawley ST, Myers RE. A randomized controlled trial of a tailored interactive computer-delivered intervention to promote colorectal cancer screening: sometimes more is just the same. Ann Behav Med. 2011 Jun;41(3):284-99. doi: 10.1007/s12160-010-9258-5. PMID 21271365
- [Background] Menon U, Belue R, Wahab S, Rugen K, Kinney AY, Maramaldi P, Wujcik D, Szalacha LA. A randomized trial comparing the effect of two phone-based interventions on colorectal cancer screening adherence. Ann Behav Med. 2011 Dec;42(3):294-303. doi: 10.1007/s12160-011-9291-z. PMID 21826576
- [Background] American Cancer Society. Cancer Facts and Figures 2014. Atlanta, GA: American Cancer Society; 2014.
- [Background] American Cancer Society. Colorectal Cancer Facts and Figures, 2014-2016. Atlanta, GA: American Cancer Society; 2014.
- [Background] Howlader N, Noone AM, Krapcho M, et al. SEER Cancer Statistics Review, 1975-2010. Bethesda, MD: National Cancer Institute, 2013.
- [Background] Edwards BK, Ward E, Kohler BA, Eheman C, Zauber AG, Anderson RN, Jemal A, Schymura MJ, Lansdorp-Vogelaar I, Seeff LC, van Ballegooijen M, Goede SL, Ries LA. Annual report to the nation on the status of cancer, 1975-2006, featuring colorectal cancer trends and impact of interventions (risk factors, screening, and treatment) to reduce future rates. Cancer. 2010 Feb 1;116(3):544-73. doi: 10.1002/cncr.24760. PMID 19998273
- [Background] Shapiro JA, Klabunde CN, Thompson TD, Nadel MR, Seeff LC, White A. Patterns of colorectal cancer test use, including CT colonography, in the 2010 National Health Interview Survey. Cancer Epidemiol Biomarkers Prev. 2012 Jun;21(6):895-904. doi: 10.1158/1055-9965.EPI-12-0192. Epub 2012 Apr 6. PMID 22490320
- [Background] Gimeno Garcia AZ, Hernandez Alvarez Buylla N, Nicolas-Perez D, Quintero E. Public awareness of colorectal cancer screening: knowledge, attitudes, and interventions for increasing screening uptake. ISRN Oncol. 2014 Mar 5;2014:425787. doi: 10.1155/2014/425787. eCollection 2014. PMID 24729896
- [Background] Gimeno Garcia AZ. Factors influencing colorectal cancer screening participation. Gastroenterol Res Pract. 2012;2012:483417. doi: 10.1155/2012/483417. Epub 2011 Dec 1. PMID 22190913
- [Background] Jepson R, Clegg A, Forbes C, Lewis R, Sowden A, Kleijnen J. The determinants of screening uptake and interventions for increasing uptake: a systematic review. Health Technol Assess. 2000;4(14):i-vii, 1-133. No abstract available. PMID 10984843
- [Background] Peterson NB, Dwyer KA, Mulvaney SA, Dietrich MS, Rothman RL. The influence of health literacy on colorectal cancer screening knowledge, beliefs and behavior. J Natl Med Assoc. 2007 Oct;99(10):1105-12. PMID 17987913
- [Background] McCaffery K, Wardle J, Waller J. Knowledge, attitudes, and behavioral intentions in relation to the early detection of colorectal cancer in the United Kingdom. Prev Med. 2003 May;36(5):525-35. doi: 10.1016/s0091-7435(03)00016-1. PMID 12689797
- [Background] Wardle J, Sutton S, Williamson S, Taylor T, McCaffery K, Cuzick J, Hart A, Atkin W. Psychosocial influences on older adults' interest in participating in bowel cancer screening. Prev Med. 2000 Oct;31(4):323-34. doi: 10.1006/pmed.2000.0725. PMID 11006057
- [Background] Robb KA, Miles A, Wardle J. Demographic and psychosocial factors associated with perceived risk for colorectal cancer. Cancer Epidemiol Biomarkers Prev. 2004 Mar;13(3):366-72. PMID 15006910
- [Background] Robb KA, Miles A, Wardle J. Perceived risk of colorectal cancer: sources of risk judgments. Cancer Epidemiol Biomarkers Prev. 2007 Apr;16(4):694-702. doi: 10.1158/1055-9965.EPI-06-0151. PMID 17416759
- [Background] Bae N, Park S, Lim S. Factors associated with adherence to fecal occult blood testing for colorectal cancer screening among adults in the Republic of Korea. Eur J Oncol Nurs. 2014 Feb;18(1):72-7. doi: 10.1016/j.ejon.2013.09.001. Epub 2013 Oct 31. PMID 24183583
- [Background] Hodge F, Maliski S, Itty T, Martinez F. Colorectal cancer screening: the role of perceived susceptibility, risk and cultural illness beliefs among American Indians. J Cult Divers. 2014 Summer;21(2):48-55. PMID 25011207
- [Background] Trauth JM, Ling BS, Weissfeld JL, Schoen RE, Hayran M. Using the transtheoretical model to stage screening behavior for colorectal cancer. Health Educ Behav. 2003 Jun;30(3):322-36. doi: 10.1177/1090198103030003007. PMID 19731499
- [Derived] Yen T, Qin F, Sundaram V, Asiimwe E, Storage T, Ladabaum U. Randomized Controlled Trial of Personalized Colorectal Cancer Risk Assessment vs Education to Promote Screening Uptake. Am J Gastroenterol. 2021 Feb 1;116(2):391-400. doi: 10.14309/ajg.0000000000000963. PMID 33009045
- See also: National Cancer Institute Colorectal Cancer Risk Assessment Tool (CCRAT) — https://ccrisktool.cancer.gov/

DOCUMENTS (2):
  • Informed Consent Form (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03819920/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03819920/Prot_SAP_002.pdf